CLINICAL TRIAL: NCT06619548
Title: The Clinical Research of Auricular Magnet for Anorexia in Children
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Responsible Party: Principal Investigator, Hung-Rong Yen, Director of the Department of Integration of Traditional Chinese-Western Medicine, China Medical University Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: CMUH112-REC1-108
Record Dates: First submitted 2024-09-27; First posted 2024-10-01 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Anorexia in Children
Keywords: anorexia in children; traditional Chinese medicine; auricular point; clinical trial

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): The participants will have auricular magnets with a strength of 1800 Gauss applied to specific acupoints in the first treatment phase. This is followed by a 14-day washout period. In the second treatment phase, the participants will have auricular magnets with no magnetic strength applied to the same acupoints.
  Interventions: Other: Auricular magnet with a magnetic strength of 1800 Gauss; Other: Auricular magnet with no magnetic strength
- Group B (Placebo Comparator): The participants will have auricular magnets with no magnetic strength applied to specific acupoints in the first treatment phase. This is followed by a 14-day washout period. In the second treatment phase, the participants will have auricular magnets with a strength of 1800 Gauss applied to the same acupoints.
  Interventions: Other: Auricular magnet with a magnetic strength of 1800 Gauss; Other: Auricular magnet with no magnetic strength

INTERVENTIONS:
Other: Auricular magnet with a magnetic strength of 1800 Gauss — Auricular magnets with a magnetic strength of 1800 Gauss are used as the experimental group.
Other: Auricular magnet with no magnetic strength — Auricular magnets with no magnetic strength are used as placebo control.

SUMMARY:
The aim of this randomized controlled cross-over trial is to explore the efficacy of auricular magnet in treating childhood anorexia. Participants will be allocated to two groups, labeled as Group A and Group B. Prior to the commencement of the trial, parents or guardians of the participants are required to fill out basic information for their children, including age, gender, height, weight, etc., and to complete the Preschooler's Eating Behavior Scale questionnaire. Over the initial 7-day period, participants of Group A receive auricular magnet therapy while participants of Group B undergo placebo magnetic auricular therapy. This is followed by a 14-day washout period to eliminate any lingering effects from the initial treatment. In the second phase, the treatments are swapped between the two groups.

DETAILED DESCRIPTION:
Anorexia in children refers to a disease in which children are not greedy for food for a long time, lose their appetite, and even refuse to eat. From the perspective of Western medicine, anorexia is classified as an eating disorder, and its causes are quite diverse, such as digestive tract diseases, neurological abnormalities, etc. From the perspective of traditional Chinese medicine (TCM), normal spleen and stomach functions are necessary for food digestion. If the spleen and stomach are not in harmony, it will cause symptoms of not breastfeeding and eating. TCM treatment of anorexia in children can be divided into two types: internal treatment and external treatment. The method of internal treatment is to give appropriate prescriptions to patients through syndrome identification and treatment. The methods of external treatment include massage, acupoint sticking, auricular point sticking, scraping therapy, navel pushing therapy, acupuncture and moxibustion, etc. Because children with anorexia do not like to eat, it is not easy to treat anorexia with drugs alone. External therapy can be considered. As traditional medicine is getting more and more attention, many patients seek TCM adjuvant treatment. This study discusses auricular point sticking in external therapy. Auricular point sticking has the advantages of noninvasiveness and convenient operation, and is suitable for children's diseases. However, the current studies on auricular points for children with anorexia are still mostly using the traditional buliuxing seeds, and there is a lack of rigorous clinical research. The aim of this study is to establish a clinical trial of auricular magnets in the treatment of anorexia in children. It is expected that subjects will be recruited from the Department of Traditional Chinese Medicine of the Affiliated Hospital of China Medical University, and the changes in eating behavior before and after treatment will be evaluated by questionnaires to explore the efficacy of auricular magnets.

ELIGIBILITY:
Inclusion Criteria:

1. The pediatric patient has one or more of the following symptoms (at least once a week and lasting for at least two months):

   1. Postprandial fullness
   2. Early satiety
   3. Epigastric pain
   4. Epigastric burning sensation or has a weight below the 15th percentile for age and sex for at least two months.
2. No prokinetic or appetite-stimulating Western medications or spleen and stomach-strengthening Chinese medications have been used within the past two weeks.

Exclusion Criteria:

Congenital abnormalities of the digestive tract, cancer, and other major illnesses, or unwillingness to cooperate with testing.

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 144 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Eating behavior change | 0, 7, 21, 28 days
  The eating behavior is evaluated by the Preschooler's Eating Behavior Scale questionnaire.

SECONDARY OUTCOMES:
Body Mass Index (BMI) change | 0, 7, 21, 28 days
  We will compare the changes in BMI values for the same patient before and after the trial to assess the effect of auricular magnets on weight.

CONTACTS AND LOCATIONS:
Overall Officials: Hung-Rong Yen, M.D., Ph.D., Study Chair — China Medical University, China
Locations (1):
- China Medical University Hospital, Taichung, Taiwan